CLINICAL TRIAL: NCT05211141
Title: Observational Study for the Evaluation of Long Term Performance and Safety of the HLS KneeTec Deep Dish Prosthesis in Total Knee Arthroplasty
Brief Title: Study to Evaluate Long Term Performance and Safety of the Knee Prosthesis (HLS KneeTec Deep Dish)
Status: Terminated | Type: Observational
Why Stopped: the clinical data collected to date is sufficient for regulatory requirements
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2017-07
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Total Knee Arthroplasty; Knee Disease; Total Knee Replacement; Osteo Arthritis Knee
Keywords: Knee Arthroplasty; Prosthesis; ultracongruent prosthesis; Implants; HLS implants; arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with knee arthroplasty: patient with HLS KneeTec Deep Dish prosthesis
  Interventions: Device: HLS KneeTec Deep Dish

INTERVENTIONS:
Device: HLS KneeTec Deep Dish — total knee arthroplasty with HLS KneeTec Deep Dish prosthesis

SUMMARY:
The aim of this study is to assess the long-term performance and safety of HLS KneeTec Deep Dish knee prosthesis when used in standard medical practice

DETAILED DESCRIPTION:
It is planned to collect prospective and retrospective data from a continuous and exhaustive series of patients in a single French site where Total Knee Arthroplasty with HLS Kneetec Deep Dish prosthesis is performed routinely

All patients treated with HLS KneeTec Deep Dish implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study.

Patients will be assessed according to the usual practice of the investigator at each participating site before surgery and then at the follow-up (FU) visits as following: 3 months (+/- 1 months); 15 months (+/- 3 months); 5 years (+/- 6 months) and 10 years (+/- 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 80 years old at the time of the surgery
* Implanted with an HLS KneeTec Deep Dish TKP according to the Instructions for Use (IFU) after the 1st of february, 2017
* Patients agree to consent to collect data from their medical records and agree to answer questionnaires for the purposes of the study.

Exclusion Criteria:

* Patients under guardianship and/or those who, according to the investigator or his delegated research team, will not be able to comply with the study procedures. (e.g. illiteracy, recent psychotic or manic disorders and/or inability to comply with routine follow-up visits.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with HLS KneeTec Deep Dish implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of implant survival in subjects receiving a total knee arthroplasty with the HLS KneeTec Deep Dish up to 10 years after the surgery | 10-year
  kaplan Meier survival rate

SECONDARY OUTCOMES:
Evaluation of functional performance of the HLS KneeTec Deep Dish after the surgery | preoperatively, 15 months, 5 years and 10 years
  International Knee Society (IKS) score
Evaluation of functional performance of the HLS KneeTec Deep Dish after the surgery | 15 months, 5 years and 10 years
  Oxford Knee Score (OKS) _ score of each question from 0 to 4 with 4 being the best outcome
Evaluation of clinical performance of the HLS KneeTec Deep Dish after the surgery | preoperatively, 15 months, 5 years and 10 years
  Devane's score_level of activity 1 to 5 with 5 being the high level of activity
Evaluation of clinical performance of the HLS KneeTec Deep Dish after the surgery | 15 months, 5 years and 10 years
  Satisfaction score on a 4-point Likert-type scale, level of satisfaction 1 to 4 with 4 being the high level of satisfaction
radiographic evaluation of the performance of HLS KneeTec Deep Dish | preoperatively up to 10 years
  component positioning
radiographic evaluation of the performance of HLS KneeTec Deep Dish | preoperatively up to 10 years
  number, severity and location of radiolucencies or osteolysis
Evaluation of safety performance during the surgery up to 10 years after the surger | starting intraoperatively up to 10-year FU
  Number, severity and casual relationship of procedure or implant-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ROCHE, MD, Principal Investigator — CHRU Nancy
Locations (1):
- Chru de Nancy, Nancy, France